CLINICAL TRIAL: NCT01280188
Title: Peroral Administration of Different Doses of Desmopressin Administered as a New Orally-Disintegrating Tablet and Desmopressin for Nasal Administration in the Treatment of CDI in Japanese Patients
Brief Title: A Study of Minirin Melt in Japanese Patients With Central Diabetes Insipidus (CDI).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE992026 CS43
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Central Diabetes Insipidus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Mellitus | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desmopressin (Experimental): Day 1 - participants continue desmopressin intranasal. Day 2 up to Day 4 - Desmopressin oral melt to optimum dose. Continue optimum dose for the four week treatment and one year follow-up periods.
  Interventions: Drug: Desmopressin Oral Melt; Drug: Desmopressin intranasal

INTERVENTIONS:
Drug: Desmopressin Oral Melt — Oral melt formulation starts on Day 2. The target initial dose of the orally disintegrating tablet is 180µg/day (60µg taken 3 times a day) and adjusted to optimally stabilise the participant's condition.
  Other Names: Minirin; FE992026
Drug: Desmopressin intranasal — Self-administered intranasal desmopressin throughout the pre-study observation period (Days -30 to Day 0) and on study Day 1

SUMMARY:
This is an open-label dose-titration study in Japanese Central Diabetes Insipidus (CDI) patients designed to demonstrate the efficacy and safety of orally-disintegrating tablet of desmopressin.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be documented to have Central Diabetes Insipidus (CDI) by at least two of the following four criteria (a-d):

  1. Failure to increase urine osmolality above 300 mOsm/kg during a period of fluid deprivation sufficient to raise plasma osmolality and sodium above the upper limit of normal level for the reference laboratory (usually 295 mOsm/kg and 148 mEq/l, respectively)
  2. Complete and continuous control of the DI by desmopressin therapy without "breakthrough" diuresis, hypernatremia, hyponatremia, or symptoms or signs of water intoxication.
  3. A deficient plasma vasopressin response to osmotic or non-osmotic stimulation.
  4. Absence of the posterior pituitary bright spot on T-1 weighted midsagittal magnetic resonance imaging (MRI) of the brain.
* Given written informed consent prior to any trial-related procedure is performed
* 24 hour urine volume (mL), urine osmolality (mOsm/kg), urine specific gravity, and serum sodium (mEq/L) maintained at a normal level by desmopressin nasal administration
* Outpatient
* The participant is, in the investigator's opinion, otherwise healthy
* Be willing and able to comply with the protocol requirements including restriction of water intake

Exclusion Criteria:

* Presence or a history of nephrogenic diabetes insipidus or diabetes mellitus
* Presence of uncorrected hypothyroidism, hypoadrenalism or hypogonadism
* Abnormalities or disease of the oral cavity that might affect the release and absorption of drug
* Unable to be placed on water-intake restriction starting from two hours before bedtime
* Presence of a hypothalamus abnormality leading to thirst disorder
* Evidence of hepatic, renal, cardiac, or pulmonary dysfunction
* Uncontrolled hypertension
* Treatment with another investigational product within the past 3 months
* Concurrent treatment with diuretics, chlorpropamide, tricyclic antidepressants, indomethacin, carbamazepine
* Alcohol dependency or drug abuse
* Breastfeeding, pregnant, or likely to become pregnant
* A mental condition, the lack of decision-making ability, dementia or a speech handicap
* Any other reason that the Investigator believes inappropriate

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in 24-hour Urine Volume | Day 0, Week 4

SECONDARY OUTCOMES:
24-hour urine volume (mL) | Day 0, Week 4
Hourly diuresis rate (mL/hr) | Day 0, Week 4
Urine osmolality (mOsm/kg) | Day 0, Week 4
Urine specific gravity (g/mL) | Day 0, Week 4
Percentage of participants within normal range for urinary output, urinary osmolality and urine specific gravity | Day 0, Week 4
Serum sodium level | up to Month 13
Participants with Adverse Events Summarized by Incidence and Severity | up to Month 13
  Includes abnormal lab values and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (5):
- Japan (5):
  - Aichi Medical University, Nagakute, Aichi, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Saitama Medical Center Jichi Medical University, Saitama, Saitama
  - Toranomon Hospital, Minato, Tokyo

REFERENCES:
- [Derived] Arima H, Oiso Y, Juul KV, Norgaard JP. Efficacy and safety of desmopressin orally disintegrating tablet in patients with central diabetes insipidus: results of a multicenter open-label dose-titration study. Endocr J. 2013;60(9):1085-94. doi: 10.1507/endocrj.ej13-0165. Epub 2013 Jun 28. PMID 23811987